CLINICAL TRIAL: NCT00291174
Title: Impedance Measurement of Epicardial Substrate for Ventricular Arrhythmias: Case Control Series of Patients With and Without Myocardial Scarring
Brief Title: Measuring Electrical Resistance of Different Tissues on the Outer Surface of the Heart
Status: Terminated | Type: Observational
Why Stopped: Unforeseen difficulty identifying and enrolling eligible subjects
Sponsor: University of Pennsylvania (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 803272
Record Dates: First submitted 2006-02-10; First posted 2006-02-13 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Cardiomyopathies; Ventricular Dysfunction; Myocardial Infarction; Arrhythmia
Keywords: Ventricular Arrhythmia; Myocardial Infarction; Ventricular Dysfunction; Coronary Artery Disease; Structural Heart Disease; Arrhythmia; Cardiomyopathies
MeSH Terms: conditions — Cardiomyopathies; Ventricular Dysfunction; Myocardial Infarction; Arrhythmias, Cardiac; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This is a research study to evaluate the electrical properties of heart tissue. The purpose of this study is to determine the impedance (electrical resistance) of different tissues on the outer surface of the heart. This may be important for distinguishing scarred heart muscle from fat that can be seen on the surface of the heart. This information may eventually be utilized in patients that undergo a procedure (called catheter ablation) for the treatment of life-threatening heart rhythms. Investigators expect a detectable difference between the impedance of normal and infarcted myocardium (approximately 50 ohms).

DETAILED DESCRIPTION:
The treatment of cardiac arrhythmias with endocardial catheter ablation has evolved rapidly over the past few decades. At the time of this writing, the ablation of almost all atrial and ventricular arrhythmias has been described in the literature. Multiple energy modalities (e.g. radiofrequency, cryotherapy) and approaches (e.g. retrograde aortic, transseptal puncture) have been described, yet ablation of some rhythms is not as successful as others.

The realization that ventricular tachycardia (VT) in the setting of Chagas Disease can originate in the epicardium has lead to the development of a percutaneous, transthoracic epicardial approach to mapping and ablation of this arrhythmia. This approach has now been applied to patients with VT in the setting of ischemic and nonischemic heart disease at many centers throughout the world. Traditional mapping technologies are utilized on the epicardium to define scarred heart tissue and locate the VT circuit.

It is well known that human hearts display a variable amount of fat overlying the epicardium. Not only is the coronary vasculature embedded in a layer of adipose tissue, but the rest of the heart may have areas of epicardial fat. As fat is an insulator and does not generate or easily conduct electrical activity, current mapping techniques may classify epicardial fat incorrectly as myocardial scar. This may have important effects on the ability to diagnose and treat arrhythmias with epicardial ablation.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients undergoing elective cardiac surgery for coronary artery disease (with or without normal heart function) or valvular disease (with normal heart function) at the Hospital of the University of Pennsylvania under the direction of Y. Joseph Woo MD will be eligible.

Exclusion Criteria:

* Patients undergoing emergent surgery and patients with idiopathic cardiomyopathy, infiltrative cardiomyopathies and hypertrophic cardiomyopathies will be excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing elective cardiac surgery for coronary artery disease
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2006-04; Primary Completion 2006-07 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J. Callans, MD, Principal Investigator — University of Pennsylvania, Dept of Medicine, Cardiology Division
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Sosa E, Scanavacca M, d'Avila A, Pilleggi F. A new technique to perform epicardial mapping in the electrophysiology laboratory. J Cardiovasc Electrophysiol. 1996 Jun;7(6):531-6. doi: 10.1111/j.1540-8167.1996.tb00559.x. PMID 8743758
- [Background] Soejima K, Stevenson WG, Sapp JL, Selwyn AP, Couper G, Epstein LM. Endocardial and epicardial radiofrequency ablation of ventricular tachycardia associated with dilated cardiomyopathy: the importance of low-voltage scars. J Am Coll Cardiol. 2004 May 19;43(10):1834-42. doi: 10.1016/j.jacc.2004.01.029. PMID 15145109
- [Background] Dixit S, Narula N, Callans DJ, Marchlinski FE. Electroanatomic mapping of human heart: epicardial fat can mimic scar. J Cardiovasc Electrophysiol. 2003 Oct;14(10):1128. doi: 10.1046/j.1540-8167.2003.03138.x. No abstract available. PMID 14521672
- [Background] Zarowitz BJ, Pilla AM. Bioelectrical impedance in clinical practice. DICP. 1989 Jul-Aug;23(7-8):548-55. doi: 10.1177/1060028089023007-803. PMID 2669371
- [Background] Casas O, Bragos R, Riu PJ, Rosell J, Tresanchez M, Warren M, Rodriguez-Sinovas A, Carreno A, Cinca J. In vivo and in situ ischemic tissue characterization using electrical impedance spectroscopy. Ann N Y Acad Sci. 1999 Apr 20;873:51-8. doi: 10.1111/j.1749-6632.1999.tb09448.x. PMID 10372149
- [Background] Cinca J, Warren M, Carreno A, Tresanchez M, Armadans L, Gomez P, Soler-Soler J. Changes in myocardial electrical impedance induced by coronary artery occlusion in pigs with and without preconditioning: correlation with local ST-segment potential and ventricular arrhythmias. Circulation. 1997 Nov 4;96(9):3079-86. doi: 10.1161/01.cir.96.9.3079. PMID 9386178
- [Background] Cinca J, Warren M, Rodriguez-Sinovas A, Tresanchez M, Carreno A, Bragos R, Casas O, Domingo A, Soler-Soler J. Passive transmission of ischemic ST segment changes in low electrical resistance myocardial infarct scar in the pig. Cardiovasc Res. 1998 Oct;40(1):103-12. doi: 10.1016/s0008-6363(98)00145-x. PMID 9876322
- [Background] Ellenby MI, Small KW, Wells RM, Hoyt DJ, Lowe JE. On-line detection of reversible myocardial ischemic injury by measurement of myocardial electrical impedance. Ann Thorac Surg. 1987 Dec;44(6):587-97. doi: 10.1016/s0003-4975(10)62141-8. PMID 3689045
- [Background] Fallert MA, Mirotznik MS, Downing SW, Savage EB, Foster KR, Josephson ME, Bogen DK. Myocardial electrical impedance mapping of ischemic sheep hearts and healing aneurysms. Circulation. 1993 Jan;87(1):199-207. doi: 10.1161/01.cir.87.1.199. PMID 8419008
- [Background] Kleber AG, Riegger CB, Janse MJ. Electrical uncoupling and increase of extracellular resistance after induction of ischemia in isolated, arterially perfused rabbit papillary muscle. Circ Res. 1987 Aug;61(2):271-9. doi: 10.1161/01.res.61.2.271. PMID 3621491
- [Background] Salazar Y, Bragos R, Casas O, Cinca J, Rosell J. Transmural versus nontransmural in situ electrical impedance spectrum for healthy, ischemic, and healed myocardium. IEEE Trans Biomed Eng. 2004 Aug;51(8):1421-7. doi: 10.1109/TBME.2004.828030. PMID 15311828
- [Background] Salazar Y, Cinca J, Rosell-Ferrer J. Effect of electrode locations and respiration in the characterization of myocardial tissue using a transcatheter impedance method. Physiol Meas. 2004 Oct;25(5):1095-103. doi: 10.1088/0967-3334/25/5/001. PMID 15535176
- [Background] Schwartzman D, Chang I, Michele JJ, Mirotznik MS, Foster KR. Electrical impedance properties of normal and chronically infarcted left ventricular myocardium. J Interv Card Electrophysiol. 1999 Oct;3(3):213-24. doi: 10.1023/a:1009887306055. PMID 10490477
- [Background] Warren M, Bragos R, Casas O, Rodriguez-Sinovas A, Rosell J, Anivarro I, Cinca J. Percutaneous electrocatheter technique for on-line detection of healed transmural myocardial infarction. Pacing Clin Electrophysiol. 2000 Aug;23(8):1283-7. doi: 10.1111/j.1540-8159.2000.tb00945.x. PMID 10962753
- [Background] Wolf T, Gepstein L, Hayam G, Zaretzky A, Shofty R, Kirshenbaum D, Uretzky G, Oron U, Ben-Haim SA. Three-dimensional endocardial impedance mapping: a new approach for myocardial infarction assessment. Am J Physiol Heart Circ Physiol. 2001 Jan;280(1):H179-88. doi: 10.1152/ajpheart.2001.280.1.H179. PMID 11123232
- [Background] Wolf T, Gepstein L, Dror U, Hayam G, Shofti R, Zaretzky A, Uretzky G, Oron U, Ben-Haim SA. Detailed endocardial mapping accurately predicts the transmural extent of myocardial infarction. J Am Coll Cardiol. 2001 May;37(6):1590-7. doi: 10.1016/s0735-1097(01)01209-8. PMID 11345370
- [Background] Zhu F, Leonard EF, Levin NW. Body composition modeling in the calf using an equivalent circuit model of multi-frequency bioimpedance analysis. Physiol Meas. 2005 Apr;26(2):S133-43. doi: 10.1088/0967-3334/26/2/013. Epub 2005 Mar 29. PMID 15798226